CLINICAL TRIAL: NCT06984640
Title: Curcumin Supplementation for the Improvement of Diabetes-related Outcomes
Acronym: CUR-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-23-7-STW; 1-503351 (Other Grant/Funding Number: Ottogi Ham Taiho Foundation)
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Over Age 60; Prediabetes or Overweight
Keywords: Curcumin; Aging
MeSH Terms: conditions — Prediabetic State; Overweight | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: * Age: Over 60 years (male and female)-preference is with pre-diabetic condition
  * Participants: around 20-25 per group (placebo and treatment)
  <Screening method>
  * Recruiting
  * Initial visit: questionnaire and fasting glucose test
    * Selecting participants: 20-25 placebo group / 20-25 curcumin supplement group
    * Criteria for selection
  * A1C level: 5.7-6.4% or
  * Fasting blood glucose level: 100-125 mg/dL
  * BMI ≥ 26-30 (≥ 30 will be considered if numbers are not enough)
    * Exclusion criteria
  * A preexisting cardiometabolic condition such as diabetes
  * Liver disease
  * Dementia
  * Tobacco use within one year prior to the study
  * Use of medications targeting diabetes or blood lipids
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin Group (Experimental): Eligible participants were randomly assigned to receive a curcumin capsule daily for 12 weeks. Each capsule contained 400 mg of a patented lipophilic matrix, delivering 80 mg of curcumin. Longvida® is a trademark of Vendure Sciences, Noblesville, IN, USA. Treatment capsules were dispensed in bottles after baseline measurements were completed, with instructions to take one capsule per day after a meal.
  Interventions: Dietary Supplement: Curcumin
- Placebo Group (Placebo Comparator): Eligible participants were randomly assigned to receive a placebo capsule daily for 12 weeks. Each capsule contained 400 mg of a patented lipophilic matrix, delivering 80 mg of dextrin with 0.05% tartrazine (a yellow food coloring). Treatment capsules were dispensed in bottles after baseline measurements were completed, with instructions to take one capsule per day after a meal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — Each capsule contained 400 mg of a patented lipophilic matrix, delivering 80 mg of curcumin. Longvida® is a trademark of Vendure Sciences, Noblesville, IN, USA.
  Arms: Curcumin Group
Dietary Supplement: Placebo — Each capsule contained 400 mg of a patented lipophilic matrix, delivering 80 mg of curcumin.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn about, test, and compare health outcomes of curcumin supplementation (400 mg). Two primary hypotheses are:

1. Curcumin supplementation will improve glycemic control in older adults with pre-diabetic conditions over a 12-week period.

   * Rationale: Curcumin has been shown to enhance insulin sensitivity, reduce fasting blood glucose, and lower HbA1c levels in preclinical and clinical studies. This hypothesis will be tested by measuring changes in fasting glucose, insulin levels, and diabetic biomarkers from baseline (Week 0) to Week 12.
2. Curcumin supplementation will beneficially alter gut microbiota composition and diversity, which is associated with improved metabolic outcomes in older adults with pre-diabetes.

   * Rationale: Curcumin is known to possess prebiotic-like properties and can influence gut microbial populations. By analyzing stool samples using metagenomic sequencing, this hypothesis will evaluate whether curcumin intake leads to increased abundance of beneficial bacteria (e.g., Akkermansia, Faecalibacterium) and decreased pathogenic taxa, alongside improved metabolic markers.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, participants were required to meet at least one of the following criteria: a) Prediabetes, defined as a fasting blood glucose level of 100-125 mg/dL or an HbA1c of 5.7-6.4%, or b) A body mass index (BMI) ≥25.

Exclusion Criteria:

* a) A preexisting cardiometabolic condition such as diabetes, b) Liver disease, c) De-mentia, d) Tobacco use within one year prior to the study, and e) Use of medications targeting diabetes or blood lipids.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Body Weight | 1 year
  Using a standard scale, body weight in kg was assessed
Body Composition | 1 year
  Using Dual-energy X-ray absorptiometry(DXA), body composition was assessed
Fat Mass Percentage | 1 year
  Using Dual-energy X-ray absorptiometry(DXA), fat mass percentage was assessed
Fat-Free Mass Percentage | 1 year
  Using Dual-energy X-ray absorptiometry(DXA), fat-free mass was assessed

SECONDARY OUTCOMES:
Triglyceride Levels | 1 year
  Blood draw followed by a Piccolo scan analyzed Triglyceride levels in the blood
Glucose Levels | 1 year
  Blood draw followed by a Piccolo scan analyzed glucose in the blood
HDL | 1 year
  Blood draw followed by a Piccolo scan analyzed HDL in the blood
LDL | 1 year
  Piccolo scan analyzed LDL in the blood
HbA1c | 1 year
  Piccolo scan analyzed HbA1c in the blood
Alanine transaminase (ALT) | 1 year
  Blood draw followed by a Piccolo scan analyzed ALT in the blood
Aspartate transaminase (AST) | 1 year
  Blood draw followed by a Piccolo scan analyzed AST in the blood

OTHER OUTCOMES:
Gut Microbiome Collection | 1 year
  Stool kits administered for fecal collection were used for gut microbiome collection

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Applied Nutrition and Exercise Science (LANES), Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided